CLINICAL TRIAL: NCT06843993
Title: A Single-Ascending Dose Clinical Trial to Study the Safety, Pharmacokinetics and Pharmacodynamics of MK-2060 in Healthy Chinese Male Adult Participants
Brief Title: Single-Ascending Dose Study of MK-2060 in Healthy Chinese Male Adult Participants (MK-2060-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 2060-009; MK-2060-009 (Other: MSD)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Panel A: MK-2060 Dose 1 (Experimental): MK-2060 dose 1 was administered as a single intravenous (IV) infusion dose on Day 1.
  Interventions: Biological: MK-2060
- Panel B: MK-2060 Dose 2 (Experimental): MK-2060 dose 2 was administered as a single IV infusion dose on Day 1. There was at least a 21-day period between dosing in Panel A and B.
  Interventions: Biological: MK-2060
- Panel C: MK-2060 Dose 3 (Experimental): MK-2060 dose 3 was administered as a single IV infusion dose on Day 1. There was at least a 21-day period between dosing in Panel B and C.
  Interventions: Biological: MK-2060
- Placebo (Placebo Comparator): Placebo was administered as a single IV infusion over MK-2060-matched time period on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MK-2060 — Single doses of MK-2060 administered via IV infusion on Day 1 according to randomization.
  Arms: Panel A: MK-2060 Dose 1; Panel B: MK-2060 Dose 2; Panel C: MK-2060 Dose 3
Biological: Placebo — Single doses of placebo administered via IV infusion on Day 1 according to randomization.
  Arms: Placebo

SUMMARY:
The goal of the study is to learn about the safety of MK-2060 and if people tolerate it. Researchers also want to learn what happens to MK-2060 in a person's body over time.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤28 kg/m^2.

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy)

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to 164 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study due to an AE | Up to 164 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who experience one or more AEs related to bleeding | Up to 164 days
  A bleeding related AE includes any sign or symptom of bleeding even if not requiring intervention by a medical/ healthcare professional, to clinically-relevant non major bleeding or major bleeding.

SECONDARY OUTCOMES:
Plasma concentration at end of infusion (Ceoi) of MK-2060 | Predose Day 1 and end of infusion
  Ceoi is defined as the amount of MK-2060 in plasma following IV infusion administration of MK-2060. Blood samples were collected at pre-specified time points to assess Ceoi.
Plasma concentration at 168 hours (C168hr) of MK-2060 | At designated timepoints (up to 168 hours)
  C168 is defined as the maximum concentration of MK-2060 reached at 168 hours postdose. Blood samples were collected at pre-specified time points to assess C168hr.
Area under the concentration versus time curve from 0 to infinity (AUC0-inf) of MK-2060 | At designated timepoints (up to 150 days)
  AUC0-inf is defined as the area under the concentration-time curve of MK-2060 from time zero to infinity. Blood samples were collected at pre-specified time points to assess AUC0-inf.
AUC from 0 to 168 hours (AUC0-168) of MK-2060 | At designated timepoints (up to 168 hours)
  AUC0-168 is defined as the area under the concentration-time curve of MK-2060 from time zero to 168 hours. Blood samples were collected at pre-specified time points to assess AUC0-168.
Time to maximum observed plasma drug concentration (Tmax) of MK-2060 | At designated timepoints (up to 150 days)
  Tmax is defined as time to the maximum concentration of MK-2060 reached. Blood samples were collected at pre-specified time points to assess Tmax.
Terminal half-life of MK-2060 | At designated timepoints (up to 150 days)
  t½ is defined as the time required to divide the MK-2060 plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-2060. Blood samples were collected at pre-specified time points to assess terminal half-life.
Clearance (CL) of MK-2060 | At designated timepoints (up to 150 days)
  CL is the volume of plasma from which MK-2060 is completely removed per unit time. Blood samples were collected at pre-specified time points to assess CL.
Volume of distribution (Vz) of MK-2060 | At designated timepoints (up to 150 days)
  Vz is defined as the distributed volume of MK-2060 in plasma. Blood samples were collected at pre-specified time points to assess Vz.
Change from baseline in activated partial thromboplastin time (aPTT) | Baseline (pre-dose) Day 1 and at designated timepoints (up to 150 days)
  Blood samples were collected at pre-specified time points to assess change from baseline in aPTT.
Anti-drug antibodies (ADA) positive incidence | At designated timepoints (up to 150 days)
  Blood samples were collected at pre-specified time points to assess the incidence of anti-MK-2060 antibodies.
Factor XI (FXI) activity level | At designated timepoints (up to 150 days)
  Blood samples were collected at pre-specified time points to assess FXI activity level.
Prothrombin time (PT) | At designated timepoints (up to 150 days)
  Blood samples were collected at pre-specified time points to assess PT.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Zhongshan Hospital,Fudan University-Dep. of Clinical Pharmacology (Site 001), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com